CLINICAL TRIAL: NCT04534049
Title: The Influence of Different Types of Physical Exercise on Immunosenescence in Elderly Persons - Senior Project Intensive Training (SPRINT)
Brief Title: The Influence of Different Types of Physical Exercise on Immunosenescence in Elderly Persons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Prof. Ivan Bautmans, Prof. dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: FRIA_SPRINT_1
Record Dates: First submitted 2020-07-03; First posted 2020-09-01 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Healthy Aged Volunteers
Keywords: Aged people; Exercises; Resistance exercise; Flexibility training; Inflammation
MeSH Terms: conditions — Motor Activity; Inflammation

ARMS (3):
- Intensive strength training (IST) (Experimental)
  Interventions: Other: Intensive Strength Training (IST)
- Strength Endurance training (SET) (Experimental)
  Interventions: Other: Strength Endurance Training (SET)
- Flexibility training (FT) (Other)
  Interventions: Other: Flexibility Training (FT)

INTERVENTIONS:
Other: Intensive Strength Training (IST)
  Arms: Intensive strength training (IST)
Other: Strength Endurance Training (SET)
  Arms: Strength Endurance training (SET)
Other: Flexibility Training (FT)
  Arms: Flexibility training (FT)

SUMMARY:
This study aims to identify the mechanisms by which physical exercise can counter inflammation and improve immune function in older persons. These mechanisms will be investigated to develop exercise-based/derived strategies to improve recovery of older patients suffering from immunosenescence and/or immune suppression.

In this randomized controlled trial, the effects of resistance exercise (RE) on inflammation and chronic low-grade inflammation (CLIP) will be investigated.

The investigators expect that exercise-induced changes in immunosenescence will be reflected by changes in the various domains of interest: 1) the expression of immunosenescence-related genes in PMBC, in circulating markers of inflammation and in PMBC behaviour following LPS stimulation, 2) the proportion of circulating PMBC showing surface and/or intracellular markers for cell senescence, and 3) markers reflecting alterations at the level of the extracellular matrix.

Additionally, the investigators want to verify whether 1) resistance exercise improves inflammation and immunosenescence in skin tissue, and 2) resistance exercise improves the stress response in skin tissue after an in-vivo inflammatory challenge by saline injection.

The results of this project will allow us to provide new insights in the complex interaction between physical exercise and immunosenescence as well as to present evidence-based guidelines for exercise in elderly persons to counter CLIP

ELIGIBILITY:
Inclusion Criteria:

* Aged people (male or female) living independently in the community;
* Aged ≥65yrs.

Exclusion Criteria:

* Performing currently or within the past six months on a regular basis physical exercise at higher intensities than habitual daily activity (e.g. fitness classes, strengthening exercises, cycling club);
* Presenting contra-indications for any of the exercise interventions;
* Cognitive impairment (unable to understand or execute the test/exercise instructions due to cognitive impairment (MMSE<24/30));
* Presenting physical disability;
* Using anti-inflammatory and/or immunosuppressive medication
* Presenting an acute inflammatory condition (CRP >10mg/L)

Exclusion Criteria for dermatology part:

* use of medications that cannot be temporarily interrupted for this study:

  * medication that suppresses allergic reaction,
  * Anticoagulation,
  * Treatment with cortisone creams, calcineurin inhibitor creams (Elidel, Protopic) within 7 days before the first visit,
  * Treatment with the following medication within 5 half-lives for the first visit: systemic immunosuppressive / immunomodulating medications (e.g. methotrexate (Ledertrexat), cyclosporine (Neoral), azathioprine (Imuran), mycomofetil phenolate (Cellcept)), Cortisone tablets (eg Medrol) (except use of cortisone in the form of nasal spray, puffer, eye drops), Targeted biological treatment (monoclonal antibodies or inhibitors, eg Dupixent),
* undergoing or have undergone allergen-specific immunotherapy,
* participating in another interventional clinical study for atopic dermatitis,
* showing inflammatory skin diseases (e.g. atopic eczema, psoriasis).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood of older adults will be investigated by qPCR to reveal changes in the inflammatory profile | Change from Baseline inflammatory profile at 6 weeks
  The primary objective is to investigate the effects of strength training on inflammation- and immunosenescence-related genes in peripheral blood mononuclear cells
Peripheral blood of older adults will be investigated by qPCR to reveal changes in the inflammatory profile | Change from Baseline inflammatory profile at 3 months
  The primary objective is to investigate the effects of strength training on inflammation- and immunosenescence-related genes in peripheral blood mononuclear cells
Peripheral blood of older adults will be investigated by qPCR to reveal changes in the inflammatory profile | Change from Baseline inflammatory profile at 6 months
  The primary objective is to investigate the effects of strength training on inflammation- and immunosenescence-related genes in peripheral blood mononuclear cells
Peripheral blood of older adults will be investigated by qPCR to reveal changes in the inflammatory profile | Change from Baseline inflammatory profile at 9 months
  The primary objective is to investigate the effects of strength training on inflammation- and immunosenescence-related genes in peripheral blood mononuclear cells
Peripheral blood of older adults will be investigated by qPCR to reveal changes in the inflammatory profile | Change from Baseline inflammatory profile at 12 months
  The primary objective is to investigate the effects of strength training on inflammation- and immunosenescence-related genes in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Jette, Brussels Capital, Belgium